CLINICAL TRIAL: NCT06047418
Title: Blepharoptosis in Indonesia: A 5-Year Retrospective Cross-Sectional Multicenter Study on Characteristics and Surgical Evaluation
Brief Title: Blepharoptosis in Indonesia: A 5-Year Multicenter Study on Characteristics and Surgical Evaluation
Status: Completed | Type: Observational
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Yunia Irawati, Director, Head of Plastic and Reconstructive Surgery Division, Department of Ophthalmology UI - RSCM, Principal Investigator, Indonesia University
Other Study IDs: 21-03-0300
Record Dates: First submitted 2023-09-14; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Blepharoptosis; Ptosis, Eyelid; Characteristics Disease; Surgical Incision
MeSH Terms: conditions — Blepharoptosis; Surgical Wound | interventions — Blepharoplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Blepharoplasty — This is an cross-sectional, retrospective observational study, to evaluate the clinical characteristics and surgical outcome of blepharoptosis patients who undergone the surgery

SUMMARY:
The goal of this observational study is to learn about blepharoptosis cases in national referral hospitals in Indonesia. The main questions it aims to answer are:

- How is the clinical characteristics, types, and surgical evaluations of blepharoptosis in this particular setting

Participant who include in this study is a patient diagnosed with blepharoptosis cases and complete medical history from January 2016 to December 2020 across 10 tertiary hospitals in Indonesia from 5 provinces

DETAILED DESCRIPTION:
The research obtained data from the medical records of 823 patients across 10 tertiary hospitals in Indonesia from 5 provinces including Cipto Mangunkusumo Hospital (Jakarta), JEC Eye Hospitals & Clinics (Jakarta), Mohammad Hoesin Hospital, Saiful Anwar Hospital, Cicendo Hospital, Sanglah Hospital, M Djamil Hospital, Wahidin Sudirohusodo Hospital, Sardjito Hospital, Kariadi Hospital, and Soetomo Hospital. Inclusion criteria entailed fully completed patient data, while exclusion criteria encompassed duplicated patient data across different years.

Patient demographic data, encompassing gender, age, and ethnicity, were extracted from the collected data. Age was divided into two groups: children (0-18 years) and adults (19-40 years, and ≥40 years). This investigation incorporated pediatric participants to assess the occurrence of blepharoptosis in children, prompted by a study revealing an 8.0% prevalence of childhood blepharoptosis.8 In age-specific relative incidence of blepharoptosis, aponeurotic and myogenic ptosis was the majority in patients younger than 40 years, emphasizing the significant association between older age and blepharoptosis prevalence, hence a cut-off of 40 years was used.7 Patient blepharoptosis classifications were established according to etiology, dividing cases into congenital and acquired categories. Acquired instances encompassed diverse etiologies (myogenic, aponeurotic, mechanical, neurogenic, traumatic, and pseudoptotic ptosis). Physical examinations discerned specific blepharoptosis traits, categorizing types as unilateral (palpebral fissure asymmetry >1 mm) and bilateral (marginal reflex distance (MRD) >2mm in both eyes).9 Levator muscle function (LF) assessment classified into excellent (≥13 mm), good (8 to 11 mm), fair (5.0 to 7 mm), and poor (≤4 mm). Severity was gauged as mild (MRD ≤2 mm), moderate (MRD 3-4mm), or severe (MRD ≥ 4mm).10 For surgical outcome evaluation, analysis depended on surgical method, success rate, and complications, divided into recurrence requiring re-operation, undercorrection, overcorrection, lagophthalmos, and asymmetry. Utilizing SPSS Statistics 25, the study employed Chi-square or Fisher's exact test and logistic regression to explore variable relationships. Initially, odds ratios were determined with bivariate analysis to examine the raw relationship between each independent variable and the outcome, without any control for other variables. Furthermore, we also computed odds ratios with multivariate analysis, which consider the simultaneous effect of multiple variables on the outcome. For this purpose, we used the stepwise method. The adequacy of our logistic regression model was assessed using the Hosmer and Lemeshow Test. A non-significant result from the Hosmer and Lemeshow Test (p>0.05) indicates that our model's predictions match the observed outcomes, suggesting that the model fits the data well.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with blepharoptosis
* complete medical record history

Exclusion Criteria:

* duplication of previously inputted cases

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: registered blepharoptosis cases from January 2016 to December 2020 across 10 tertiary hospitals in Indonesia from 5 provinces, including Cipto Mangunkusumo Hospital (Jakarta), JEC Eye Hospitals & Clinics (Jakarta), Mohammad Hoesin Hospital, Saiful Anwar Hospital, Cicendo Hospital, Sanglah Hospital, M Djamil Hospital, Wahidin Sudirohusudo Hospital, Sardjito Hospital, Kariadi Hospital, and Soetomo Hospital
Sampling Method: Probability Sample
Enrollment: 823 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-04-07 (Actual); Study Completion 2023-08-03 (Actual)

PRIMARY OUTCOMES:
Demographic and Clinical Characteristic | 2021-2022
  demographics were categorised into sex, age and race while clinical characteristic were including type of ptosis, laterality, mechanism, severity, elevator function. we use percentage to calculate the proportion of the patients
Surgical technique | 2021-2022
  we collect the data history of patient's eyes who were undergoing the surgery. we use percentage to calculate the proportion of each surgical technique used as frontal suspension, levator resection, elevator advancement, fasanella servant, mullerectomy and tumor excision

SECONDARY OUTCOMES:
surgical evaluations | 2021-2022
  surgical evaluations were observed and calculated from the current complications appeared in percentage

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto Mangunkusumo Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided
It depends on what is the aim of the research, and we should collaborate to do the research